CLINICAL TRIAL: NCT05184361
Title: Effects of Intermittent Versus Continuous Energy Restriction on Metabolic Adaptation in Women With Obesity
Acronym: BREAK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: University of Lisbon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BREAKSTUDY2021
Record Dates: First submitted 2021-12-17; First posted 2022-01-11 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Obesity; Weight Loss
Keywords: Adaptive Thermogenesis; Metabolic Slowing
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent energy restriction (IER) (Experimental): Initially participants will undergo 2-weeks of neutral energy balance (EB). After this, the IER will consist of: 2-weeks of energy restriction interspersed with 1-week in neutral EB (total of 23-week period).
  At the end, 8-weeks in neutral EB will be required.
  Interventions: Behavioral: Intermittent energy restriction (IER)
- Continuous energy restriction (CER) (Active Comparator): Similarly to IER, CER participants will undergo 2-weeks of neutral EB. After this, the CER will consist of: 16-weeks of continuous energy restriction. At the end, 8-weeks in neutral EB will be required.
  Interventions: Behavioral: Continuous energy restriction (CER)

INTERVENTIONS:
Behavioral: Intermittent energy restriction (IER) — Both groups will be accompanied by a registered dietitian in order to provide an individual and personalized diet plan that will suppress the respective daily requirements for each phase. Macronutrient distribution will be the following: 35% protein, 35% carbohydrate and 30% fat.
  Daily energy requirements (DER) will be calculated by multiplying measured RMR (through indirect calorimetry) by physical activity level (PAL), assessed by accelerometry.
  In order to achieve a neutral EB, 100% of their daily energy requirements (DER) will be prescribed for each participant. For both groups, an energy restriction of 33% of one's DER will be created. The IER group will alternate between 2-weeks in energy restriction (67% DER) and 1-week in neutral EB (100% DER), in a total of 23-weeks.
  The IER group will alternate between 2-weeks in energy restriction (67% DER) and 1-week in neutral EB (100% DER), in a total of 23-weeks.
  Arms: Intermittent energy restriction (IER)
Behavioral: Continuous energy restriction (CER) — A dietary plan comprising 67% of DER will be prescribed to the CER group. Participants will be asked to follow this plan in a total of 16-weeks, without interruptions.
  Arms: Continuous energy restriction (CER)

SUMMARY:
One of the major challenges for treating obesity is to maintain a weight reduced state on the long term due to the high rate of weight regain. Therefore, the aim of this study is to evaluate the effects of an intermittent versus a continuous energy restriction in body composition (body weight, fat mass and fat-free mass) and metabolic adaptation, in women with obesity.

DETAILED DESCRIPTION:
Literature is full of lifestyle interventions aimed for weight loss (WL) in several populations. However, one of the major challenges for treating obesity is WL maintenance on the long term due to the high rate of weight regain.

The reduction of the resting metabolic rate (RMR) is one of the identified aspects regarding compensatory metabolic alterations. After a WL intervention, decreases in RMR are mainly explained by the loss of fat-mass (FM) and fat-free mass (FFM). However, some authors showed that these reductions tend to be higher than predicted (explained by FM and FFM loss), a phenomenon called "metabolic adaptation" (MA). MA has been studied as a possible barrier to WL, WL maintenance and may contribute to weight regain. However, its relevance on long-term WM has been recently questioned. It is known that in order to lose weight, a negative energy balance (EB) must be achieved, meaning when EE surpasses the energy intake (EI). However, this negative EB may be achieved through several strategies, by changing the EI (energy restriction (ER)) and/or EE (increasing physical activity).

Regarding EI strategies, continuous energy restriction (CER) is the most common nutritional strategy for WL, consisting in a daily energy restriction according to one's specific needs. However, some concern has been pointed out regarding this widely used strategy, once it evolves several behavioural, metabolic and endocrine responses that may contribute to therapeutic adherence, undermining WL and its maintenance. On the other hand, intermittent energy restriction (IER) has been recently suggested as an alternative to CER. IER consists in interspersing periods of ER with periods of neutral EB, called "refeed" or "diet breaks" during the WL phase. Energy restriction is followed by several adaptive responses, namely endocrine, including thyroid, appetite regulation and steroid hormones, influencing the energy expenditure (EE), body composition and satiety. Therefore, understanding how hormones may influence RMR and as a consequence, AT, it´s crucial to a better understanding.

According to the literature, compensatory metabolic responses following ER and WL can be reversed following a 7-to-14-day period of energy balance post-weight loss. Therefore, considering that the length of the nutritional intervention for WL may benefit a reduction, we consider relevant to study other ER designs/patterns, namely 2 weeks in ER interspersed with 1 week in EB, comparing to a CER. Taking into account this therapeutic as a potential opportunity for the obesity's treatment, this paper describes the protocol for a randomized controlled trial (RCT), which targets to evaluate the effects of an IER (alternating 2 weeks of ER with 1 in neutral EB), comparing to a CER. This trial aims: a) to compare the effects of a IER vs CER strategy on body composition variables (body weight, fat mass and fat-free mass) and in metabolic adaptation and, b) to understand if participants will be able to maintain a reduced weight state after 12 months (successful weight-loss maintenance), in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Women
* BMI ranging between 30 and 39.9 kg/m2
* Age between 20-45 years
* Weight stable in the last 6 months (less than 5% weigh variation)
* Inactive (less then 150 min/week of moderate physical activity or 75 min/week of vigorous physical activity
* Living in Lisbon Metropolitan Area and being able to drive to Faculty of Human Kinetics and Germano de Sousa Laboratory (Algés)
* Available to be randomized to any of the trial groups (CER or IER)
* Willing to commit with the assigned group protocol, including the nutritional intervention and lifestyle recommendations, as well as being available for participation in all evaluation moments.

Exclusion Criteria:

* Previous or present health disorders: cancer, autoimmune, cardiac, psychiatric, kidney and liver disease (except liver steatosis), diabetes, chronic intestinal inflammatory disease, or other medical conditions known to affect energy balance homeostasis
* Menopause
* Hormonal or thyroid disorder
* Medications that promote weight gain or alter energy balance, including corticosteroids, antidepressants, anxiolytics, mood-stabilizing, and antipsychotics
* Medications or dietary supplements for weight-loss in the past 3 months
* Pregnant for the past 6 months or breastfeeding
* Planning to get pregnant in the next 2 years or getting pregnant during the study
* Current consumption of more than 14 alcoholic drinks per week or other substance abuse, and/or current acute treatment or rehabilitation program for alcohol/substance abuse
* Surgery or in hospital admission for the last month
* Positive for Covid-19 in the past 3 months or testing positive during the intervention phase of the study

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Fat mass | 24 months
  To estimate total fat mass (FM), dual energy X-ray absorptiometry (Hologic Explorer-W, Waltham, USA) will be used. A whole-body scan will be performed and the attenuation of X-rays pulsed between 70 and 140 kV synchronously with the line frequency for each pixel of the scanned image will be measured.
Adaptive thermogenesis (AT) | 24 months
  AT will be assessed as: AT (kcal/d) = (pREE at the end of the intervention - mREE at the end of the intervention) - (pREE baseline - mREE baseline)

SECONDARY OUTCOMES:
Weight | 24 months
  Weight will be determined using a digital scale, with 0,1 kg interval (Seca, Hamburg, Germany).
Height | Baseline
  Height will be determined using a stadiometer Seca 704 s, with 0,1 cm intervals (Seca, Hamburg, Germany)
Body mass index (BMI) | 24 months
  BMI will be calculated using the formula [weight (kg)/height2(m2)]
Fat-free mass (FFM) | 24 months
  To estimate fat-free mass (FFM), dual energy X-ray absorptiometry (Hologic Explorer-W, Waltham, USA) will be used. A whole-body scan will be performed and the attenuation of X-rays pulsed between 70 and 140 kV synchronously with the line frequency for each pixel of the scanned image will be measured.
Resting energy expenditure (REE) | 24 months
  REE will be determined using indirect calorimetry COSMED Fitmate device (Cosmed, Rome, Italy) will be used to measure breath-by-breath oxygen consumption (V̇O2 ) and carbon dioxide production (V̇CO2) using a facial mask.
Energy balance (EB) | 24 months
  The EB will be calculated as: EB (kcal/d) = 1.0 * (ΔFMM/Δt) + 9.5 * (ΔFM/Δt). ΔFM and ΔFFM represent the change in grams of FM and FFM from the beginning to end of the intervention and Δt is the time length of the intervention in days.
Free-living physical activity | 24 months
  The amount of activity assessed by the Actigraph accelerometer will be expressed as minutes per day spent in different intensities. The cutoff values used to define the intensity of PA and therefore to quantify the mean time in each intensity (sedentary, light, moderate or vigorous) will be: sedentary: < 100 counts·min-1; light: 100-2019 counts·min-1; moderate: 2020-5998 counts·min-1 (corresponding to 3-5.9 METs); vigorous: ≥ 5999 counts·min-1 (corresponding to ≥6 METs). A valid day will be defined as having 600 or more minutes (≥10h) of monitor wear during waking hours.
Total daily energy expenditure (TDEE) | 24 months
  TDEE will be assessed by the Actigraph accelerometer using the Crouter et al equations.
Physical activity energy expenditure (PAEE) | 24 months
  PAEE will be calculated as total energy expenditure (TEE) minus (0.1*TEE + REE), assuming the thermic effect of food represents 10% of TEE, and REE represents Resting energy expenditure.
Blood thyroid levels | 24 months
  Free T3 and free T4 will be run by immunoassay with chemiluminescent detection (Advia Centaur, Siemens).
Blood insulin levels | 24 months
  Blood insulin levels assessment will be performed in an automated analyser with chemiluminescent detection [Advia Centaur, Siemens].
Blood leptin levels | 24 months
  Serum levels of leptin will be measured by enzyme immunoassay [ELISA].
Blood cortisol levels | 24 months
  Blood levels of cortisol will be determined by immunoassay with chemiluminescence detection [Advia Centaur, Siemens].

CONTACTS AND LOCATIONS:
Overall Officials: Vítor H Teixeira, PhD, Principal Investigator — Faculty of Nutrition and Food Sciences, University of Porto; Analiza M Silva, PhD, Principal Investigator — Faculty of Human Kinetics, University of Lisbon
Locations (1):
- Faculdade de Motricidade Humana da Universidade de Lisboa, Cruz Quebrada, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cortez FM, Nunes CL, Sardinha LB, Silva AM, Teixeira VH. The BREAK study protocol: Effects of intermittent energy restriction on adaptive thermogenesis during weight loss and its maintenance. PLoS One. 2023 Nov 13;18(11):e0294131. doi: 10.1371/journal.pone.0294131. eCollection 2023. PMID 37956119